CLINICAL TRIAL: NCT03056573
Title: Assessment of the St Jude Medical Portico Resheathable Aortic Valve System-Alternative Access
Acronym: Portico ALT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJM-CIP-10144
Record Dates: First submitted 2017-01-31; First posted 2017-02-17 (Actual); Results first posted 2020-03-17 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVI; Valvular heart disease; Transcatheter aortic valve implantation
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: Portico TF and ALT Delivery System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subclavian/axillary (Experimental): Subclavian/axillary access route
  Interventions: Device: Subclavian /Axillary TAVR implant
- Transaortic (Experimental): Transaortic access route
  Interventions: Device: Transaortic TAVR Implant

INTERVENTIONS:
Device: Transaortic TAVR Implant — Transaortic TAVR implant
  Arms: Transaortic
Device: Subclavian /Axillary TAVR implant — Subclavian /Axillary TAVR implant
  Arms: Subclavian/axillary

SUMMARY:
Expand the indication of the Portico TF Delivery System and obtain approval of the Alternative Access Delivery System

DETAILED DESCRIPTION:
Expand the indication of the Portico TF Delivery System and obtain approval of the Alternative Access Delivery System to place a Portico transcatheter aortic valve through an alternative access site, specifically subclavian/axillary or transaortic (TAo) in subjects with symptomatic severe native aortic stenosis who are considered high surgical risk

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent prior to uploading CT scan to core lab.
2. Subject is ≥ 18 years of age or legal age in host country.
3. Subject's aortic annulus diameter meets the range indicated in the Instructions for Use as measured by multislice CT conducted within 180 days prior to the index procedure.
4. Subject has senile degenerative aortic stenosis seen by echocardiography within 90 days of index procedure as measured by:

   1. mean gradient >40 mmHg
   2. Peak velocity ≥ 4.0 m/s
   3. Doppler Velocity Index <0.25
   4. Aortic valve area (AVA) of ≤ 1.0 cm2 or indexed EOA ≤ 0.6 cm2/m2).
5. Subject has symptomatic aortic stenosis as demonstrated by NYHA Functional Classification of Class II, or greater or other symptoms of aortic stenosis (e.g. syncope).
6. Subject is deemed high operable risk and preferred TAVI delivery route is alternate access (subclavian/axillary or direct aortic) per the medical opinion of the center's heart team and confirmed by SSC.

   * High risk is defined as an STS mortality > 8% or documented heart team agreement ≥ high risk for SAVR due to frailty or co-morbidities

Exclusion Criteria:

1. Subject is unwilling or unable to comply with all study-required follow-up evaluations.
2. Subject has a documented history of a cerebral vascular accident (CVA) or transient ischemic attack (TIA) within 6 months (less than or equal to 180 days) prior to the index procedure.
3. Subject has carotid artery disease requiring intervention.
4. Subject has evidence of a myocardial infarction (MI) within 30 days prior to patient index procedure.
5. Subject has a native aortic valve that is congenitally unicuspid, bicuspid, quadricuspid or non-calcified as seen by echocardiography.
6. Subject has severe mitral valvular regurgitation.
7. Subject has severe mitral stenosis.
8. Subject has a pre-existing prosthetic cardiac device, valve, or prosthetic ring in any position.
9. Subject refuses any blood product transfusion.
10. Subject has resting left ventricular ejection fraction (LVEF) less than 20%.
11. Subject has documented, untreated symptomatic coronary artery disease (CAD) requiring revascularization.
12. Subject has had a percutaneous interventional or other invasive cardiovascular or peripheral vascular procedure less than or equal to 14 days prior to index procedure.
13. Subject has severe basal septal hypertrophy that would interfere with transcatheter aortic valve placement.
14. Subject has a history of, or is currently diagnosed with, endocarditis.
15. There is imaging evidence of intracardiac mass, thrombus, or vegetation.
16. Subject is considered hemodynamically unstable (requiring inotropic support or mechanical heart assistance).
17. Subject is in acute pulmonary edema or requiring intravenous diuretic therapy to stabilize heart failure.
18. Subject with severe pulmonary disease as determined by STS score.
19. Subject is on chronic oral steroid therapy.
20. Subject has a documented hypersensitivity or contraindication to anticoagulant or antiplatelet medication.
21. Subject has renal insufficiency as evidenced by a serum creatinine greater than 3.0 mg/dL (265.5 µmol/L) or end-stage renal disease requiring chronic dialysis.
22. Subject has morbid obesity defined as a BMI greater than or equal to 40.
23. Subject has ongoing infection or sepsis.
24. Subject has uncontrolled blood dyscrasias as defined: leukopenia (WBC<3000 mm3), acute anemia (Hb<9 mg/dL), thrombocytopenia (platelet count <50,000 cells/mm3,).
25. Anatomy falling outside the recommended values in the IFU, unless specifically approved by the Subject Selection Committee.
26. Subject has an active peptic ulcer or has had gastrointestinal (GI) bleeding within 90 days prior to the index procedure.
27. Subject is currently participating in another investigational drug or device study, unless approved by the Sponsor.
28. Subject has/had emergency surgery for any reason within 30 days of the index procedure.
29. Subject has a life expectancy less than 1 year.
30. Subject has other medical, social or psychological conditions that, in the opinion of the Principal Investigator or the Subject Selection Committee, preclude the subject from study participation.
31. Subject is diagnosed with a state of dementia which would fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits.
32. Subject has a documented allergy to contrast media that cannot adequately be treated, nitinol alloys, porcine tissue, or bovine tissue.
33. Significant aortic disease including abdominal aortic or thoracic aneurysm defined as maximal luminal diameter 5cm or greater
34. Subjects with severe pulmonary hypertension and severe RV dysfunction
35. Subjects with hypertrophic cardiomyopathy

Transaortic Subject Cohort Specific Exclusion Criteria

Subjects are not eligible for participation in the TAo access arm if they meet any of the following exclusion criteria:

1. Subject has a chest condition (anatomical or otherwise) that prevents TAo access.
2. Subject has pre-existing patent RIMA graft that would preclude access.
3. Subject has a porcelain aorta, defined as an extensive circumferential calcification of the ascending aorta that would complicate TAo access.

Subclavian/Axillary Subject Cohort Specific Exclusion Criteria

Subjects are not eligible for participation in the subclavian/axillary access arm if they meet any of the following exclusion criteria:

1. Subject's access vessel (subclavian/axillary) diameter will not allow for introduction of the 18/19 Fr delivery system.
2. Subject's subclavian/axillary arteries have severe calcification and/or tortuosity.
3. Subject has a history of LIMA/RIMA graft that would preclude access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-07-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Rigshospitalet Copenhagen, Copenhagen, Denmark
- Germany (3):
  - Deutsches Herzzentrum Berlin, Berlin
  - Herzzentrum Leipzig GmbH, Leipzig
  - Universitatsklinikum Tubingen Medizinische Klinik-Kardio, Tübingen
- Italy (2):
  - Ospedale Niguarda Ca'Granda, Milan
  - Policlinico San Donato, San Donato Milanese
- Netherlands (3):
  - Amsterdam Academic Medical Centre (AMC), Amsterdam
  - Medical Center Leeuwarden, Leeuwarden
  - UMC St Radboud, Nijmegen
- Basel University Hospital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Wely M, Bruschi G, Bedogni F, Thiele H, Jeger RV, van der Wulp K, Soendergaard L, Kempfert J, Schlensak C, Linke A. Clinical Outcomes of the Portico Transcatheter Aortic Valve Delivered via Alternative Access: 30-Day and 1-Year Results of the Portico ALT Study. J Invasive Cardiol. 2020 Nov;32(11):405-411. doi: 10.25270/jic/20.00109. Epub 2020 Aug 10. PMID 32771997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 64 subjects were enrolled and undergone implant with a Portico Transcatheter Aortic Valve via an alternative access route at 10 sites between March 29, 2017 and June 04, 2018.
Pre-assignment Details: Of the 64 subjects, 45 subjects were implanted via subclavian/axillary access and 19 via transaortic access. Enrollment in the transaortic arm was stopped after 15 months due to a slow enrollment rate. All subjects will be followed through 1-year post implant.
Groups:
- Subclavian/Axillary Access Arm: Subjects who underwent TAVR with the Portico THV via the subclavian or axillary alternative access site.
- Transaortic Access Arm: Subjects who underwent Transaortic TAVR implant.
Period: Overall Study
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Started | 45 | 19
Completed | 40 | 14
Not Completed | 5 | 5
Not completed — Death | 2 | 4
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Transaortic Arm: Subjects who underwent Transaortic TAVR implant.
- Total: Total of all reporting groups
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Arm | Total
Number analyzed (Participants) | 45 | 19 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.7 (5.9) | 77.1 (7.2) | 80.3 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 10 | 36
  Male | 19 | 9 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 45 | 19 | 64
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 14 | 3 | 17
  Switzerland | 2 | 0 | 2
  Germany | 5 | 3 | 8
  Denmark | 1 | 0 | 1
  Netherlands | 23 | 13 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Vascular Complications
Description: Major Vascular complication is defined as
  * Any aortic dissection, aortic rupture, annulus rupture, left ventricle perforation, or new apical aneurysm/pseudo-aneurysm or
  * Access site or access-related vascular injury leading to death, life-threatening or major bleeding, visceral ischaemia or neurological impairment or
  * Distal embolization from a vascular source requiring surgery or resulting in amputation or irreversible end-organ damage or
  * The use of unplanned endovascular or surgical intervention associated with death, major bleeding, visceral ischaemia or neurological impairment or
  * Any new ipsilateral lower extremity ischemia documented by patient symptoms, physical exam, and/or decreased or absent blood flow on lower extremity angiogram or
  * Surgery for access site-related nerve injury or
  * Permanent access site-related nerve injury
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 45 | 19
Participants | 2 | 1

2. Secondary Outcome: Number of All- Cause Mortality
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 45 | 19
Participants | 1 | 2

3. Secondary Outcome: Number of All- Cause Mortality
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 45 | 19
Participants | 2 | 4

4. Secondary Outcome: Cardiovascular Mortality
Description: Any 1 of the following criteria:
  * Death due to proximate cardiac cause (e.g., myocardial infarction, cardiac tamponade, worsening heart failure)
  * Death caused by non-coronary vascular conditions such as neurological events, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular disease.
  * All procedure-related deaths, including those related to a complication of the procedure or treatment for a complication of the procedure
  * All valve-related deaths including structural or nonstructural valve dysfunction or other valve-related adverse events
  * Sudden or unwitnessed death
  * Death of unknown cause
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 45 | 19
Participants | 0 | 2

5. Secondary Outcome: Cardiovascular Mortality
Description: as for outcome 4
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 45 | 19
Participants | 1 | 4

6. Secondary Outcome: Number of Participants With Disabling Stroke
Description: Disabling stroke is an mRS score of 2 or more at 90 days and an increase of at least 1 mRS category from an individual's prestroke baseline
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 45 | 19
Participants | 1 | 0

7. Secondary Outcome: Number of Participants With Disabling Stroke
Description: as for outcome 6
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 45 | 19
Participants | 1 | 0

8. Secondary Outcome: Number of Participants With Non-disabling Strokes
Description: Non-disabling is an mRS score of <2 at 90 days or 1 that does not result in an increase of at least 1 mRS category from an individual's prestroke baseline
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 45 | 19
Participants | 4 | 0

9. Secondary Outcome: Number of Participants With Non-disabling Strokes
Description: as for outcome 8
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 45 | 19
Participants | 4 | 0

10. Secondary Outcome: Number of Participants With Life Threatening Bleeding Requiring Transfusion
Description: Life threatening bleeding requiring transfusion
  * Overt bleeding either associated with a drop in the hemoglobin level of at least 3.0 g/dL or requiring transfusion of 2 or 3 units of whole blood/RBC, or causing hospitalization or permanent injury, or requiring surgery AND
  * Does not meet criteria of life-threatening or disabling bleeding
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 45 | 19
Participants | 2 | 2

11. Secondary Outcome: Number of Participants With Life Threatening Bleeding Requiring Transfusion
Description: as for outcome 10
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 45 | 19
Participants | 2 | 2

12. Secondary Outcome: Number of Participants With Acute Kidney Injury Requiring Dialysis
Description: Increase in serum creatinine to greater than or equal to 300% (3 X increase compared with baseline) or serum creatinine of ≥ 4.0 mg/dL (354 mmol/L) with an acute increase of at least 0.5 mg/dL (44 mmol/L)or Urine output <0.3 mL/kg per hour for ≥24 hours or anuria for ≥12 hours. Patients receiving renal replacement therapy are considered to meet Stage 3 criteria irrespective of other criteria
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 45 | 19
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Acute Kidney Injury Requiring Dialysis
Description: as for outcome 12
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 45 | 19
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With Composite of Periprocedural Encephalopathy, All Stroke and All TIA
Description: Stroke is an acute symptomatic episode of neurological dysfunction attributed to a vascular cause.
  Transient Ischemic Attack (TIA) is a transient (less than 24 hrs) episode of neurological dysfunction caused by focal brain, spinal cord, or retinal ischemia, without acute infarction. No evidence of infarction if imaging performed.
  Encephalopathy is defined as altered mental state (e.g., seizures, delirium, confusion, hallucinations, dementia, coma, psychiatric episode).
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 45 | 19
Participants | 5 | 0

15. Secondary Outcome: Number of Participants With Composite of Periprocedural Encephalopathy, All Stroke and All TIA
Description: as for outcome 14
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 45 | 19
Participants | 5 | 0

16. Secondary Outcome: Number of Participants With Moderate and Severe Aortic Regurgitation
Time Frame: 1 year
Population: The number of participants who were available at that time point were included
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 28 | 13
Participants | 1 | 1

17. Secondary Outcome: Change in NYHA Class From Baseline to 30 Days
Description: New York Heart Association (NYHA) functional classification provides a way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina pain.
  Class I. Patients with cardiac disease but without resulting limitation of physical activity.
  Class II. Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest.
  Class III. Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest.
  Class IV. Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest.
Time Frame: Baseline to 30 days
Population: We had presented the data only for the participants who had an outcome at baseline and at 30 days (paired data).
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 40 | 13
Participants
  Improvement from Baseline (BL) NYHA I to 30days | 0 | 0
  Improvement from BL NYHA II to 30days NYHA I | 3 | 2
  Improvement from BL NYHA III to 30days NYHA I & II | 25 | 8
  Improvement fromBL NYHA IV to 30days NYHA I,II,III | 3 | 0

18. Secondary Outcome: Change in Six Minute Walk Test From Baseline as Compared to 30 Days
Description: The Six Minute Walk Test (6MWT)measures the distance that a patient can walk in a period of 6 minutes. The distance walked is measured in meters. This test measures the patients' functional status. The more meters a patient can walk over baseline indicates improvement in functional status.
Time Frame: Baseline to 30 days
Population: We had presented the data only for the participants who had an outcome at baseline and at 30 days (paired data).
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 39 | 9
Meter | 46.3 (94.7) | 6.0 (87.3)

19. Secondary Outcome: Change in Effective Orifice Area From Baseline as Compared to 30 Days
Description: Effective Orifice Area of the prosthetic valve measured via echocardiography to determine physiological area of blood flow through the valve.
Time Frame: Baseline to 30 days.
Population: We had presented the data only for the participants who had an outcome at baseline and at 30 days (paired data).
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 20 | 8
cm2 | 1.1 (0.3) | 1.0 (0.3)

20. Secondary Outcome: Number of Participants With Overall Acute Device Success
Description: Acute device success is defined as a subject who achieves a) successful vascular access, delivery and deployment of the device and successful retrieval of the delivery system, b) correct position of the device in the proper anatomical location, c) intended performance of the prosthetic heart valve, and d) only 1 valve implanted in the proper anatomical location.
  Device success is a 'technical' composite endpoint meant to characterize the acute device and procedural factors which underlie vascular access, delivery, and performance of the TAVI system. Echocardiography should be routinely utilized as the standard for measuring prosthetic valve stenosis and regurgitation immediately after TAVI, and should always be performed in a resting state, either within 24-48 h after the index procedure or before hospital discharge.
Time Frame: 7 days
Population: The number of participants who were available at that time point were included
Measure: Count of Participants; unit: Participants
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
Number analyzed (Participants) | 45 | 16
Participants | 43 | 14

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Subclavian/Axillary Access Arm | Transaortic Access Arm
All-Cause Mortality (participants affected / at risk) | 2/45 | 4/19
Serious Adverse Events (participants affected / at risk) | 21/45 | 15/19
Other Adverse Events (participants affected / at risk) | 30/45 | 9/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subclavian/Axillary Access Arm (N=45) | Transaortic Access Arm (N=19)
Anemia (Blood and lymphatic system disorders) | 2 | 1
Chronic Lymphedema (Blood and lymphatic system disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 1
Cardiac Arrhythmias (Cardiac disorders) | 0 | 1
Complete Heart Block (Cardiac disorders) | 1 | 1
Heart Failure (Cardiac disorders) | 1 | 1
Left Bundle Branch Block (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 1
Pericardial Tamponade (Cardiac disorders) | 0 | 1
Sick Sinus Syndrome (Cardiac disorders) | 1 | 0
GI Bleed (Gastrointestinal disorders) | 2 | 0
Death of unknown cause (General disorders) | 1 | 2
Increasing Pain On Both Legs (General disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Fever (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 3
Sepsis (Infections and infestations) | 1 | 0
Access Site Bleeding Event (Injury, poisoning and procedural complications) | 1 | 0
Broken Arm Right Side (Injury, poisoning and procedural complications) | 1 | 0
Broken Left Leg (Injury, poisoning and procedural complications) | 1 | 0
Broken Leg With Hospitalization (Injury, poisoning and procedural complications) | 1 | 0
Cardiac Perforation (Injury, poisoning and procedural complications) | 0 | 1
Femoral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Re-Fracture Left Leg (Injury, poisoning and procedural complications) | 1 | 0
Vascular Access Site and Access Related Complications (Injury, poisoning and procedural complications) | 1 | 0
Stroke (Nervous system disorders) | 4 | 0
Transient Ischemic Attack (TIA) (Nervous system disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Device Embolization (Surgical and medical procedures) | 1 | 0
Vessel Dissection (Surgical and medical procedures) | 2 | 0
Bleeding (Vascular disorders) | 3 | 2
Reduced Left Ventricular Function/ Subclinical Heart Failure (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subclavian/Axillary Access Arm (N=45) | Transaortic Access Arm (N=19)
Access Site Bleeding Event (Injury, poisoning and procedural complications) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 3
Atrial Fibrillation (Cardiac disorders) | 4 | 1
Bleeding (Vascular disorders) | 6 | 1
Complete Heart Block (Cardiac disorders) | 2 | 0
Congestive Heart Failure (Cardiac disorders) | 2 | 0
First Degree Heart Block (Cardiac disorders) | 4 | 2
Hematoma (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 3 | 0
Left Bundle Branch Block (Cardiac disorders) | 9 | 1
Pseudoaneurysm (Vascular disorders) | 2 | 0
Right Bundle Branch Block (Cardiac disorders) | 2 | 0
Vessel Dissection (Injury, poisoning and procedural complications) | 5 | 0
Accelerated Junctional Rhythm (Cardiac disorders) | 1 | 0
Delirium (Nervous system disorders) | 2 | 0
Mild Congestive Heart Failure (Cardiac disorders) | 1 | 0
Pain Shoulder Left Access Site Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Painful Left Arm (With Impaired Mobility) (Musculoskeletal and connective tissue disorders) | 1 | 0
Painful Right Groin (Diagnostic Site) (Injury, poisoning and procedural complications) | 1 | 0
Pinched Nerve (Injury, poisoning and procedural complications) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Supraventricular Extrasystole (Cardiac disorders) | 1 | 1
Transient LBBB (Cardiac disorders) | 1 | 0
Ventricular Extrasystole (Cardiac disorders) | 1 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1
Infection (Infections and infestations) | 0 | 1
Renal Insufficiency/Worsening Renal Function (Renal and urinary disorders) | 0 | 1
Ventricular Fibrillation (Cardiac disorders) | 0 | 1
Left Anterior Fascicular Block (Cardiac disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 2 | 0
Ankle Edema (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Dizziness And Short-Term Disorientation (General disorders) | 1 | 0
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Syncope Epileptic Insult (Nervous system disorders) | 1 | 0
Aortic Valve Stenosis (Cardiac disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT03056573/Prot_SAP_000.pdf